CLINICAL TRIAL: NCT06986694
Title: Effects of Voodoo Flossing Technique on Pain, Range of Motion and Physical Function in Patients With Knee Osteoarthritis: A Randomized Control Study
Brief Title: Effects of Voodoo Flossing Technique in Knee Osteoarthritis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0153
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthritis; Pain; Range of Motion; Physiotherapy
Keywords: Knee Osteoarthritis; Pain; Physical Function; Physiotherapy; Range of Motion; Voodoo Flossing
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Voodoo Flossing technique along with aerobic & strengthening exercises and conventional protocol. (Experimental): Patient will sit or lie down comfortably with affected knee exposed and in extension. Start by wrapping voodoo floss band at the shin bone just below the knee joint with 50% tension in the band and 50% overlapping on each wrap by working your way up towards the thigh. Keep the flossing band on for at least 1-2 minutes and perform gentle knee movements to promote mobility.
  * Knee flexion and extension in full range of motion in standing position 20-30 sec.
  * Knee squats with/without support 20-30 sec.
  * Abduction and Adduction 20-30 sec. Perform each exercise with 10-15 seconds of rest between each set. After completing ROM exercises, allow the knee to rest in comfortable position and then carefully unwrap the voodoo band from the knee joint. Also monitor the knee for any changes.
  Interventions: Other: Group A will receive Voodoo Flossing Technique along with aerobic and strengthening exercises & conventional physiotherapy protocol for Knee OA.
- Aerobic and strength training and conventional physiotherapy protocol for knee OA. (Active Comparator): Aerobic Exercises: Walking or Stationary Cycling 2 times a week for 4 weeks. Walking: On flat surface or Treadmill 10 minutes warm-up, 30 minutes brisk walking, 5 minutes cool down. Cycling: Ergometer cycling
  * 10 minutes warm-up, 30 minutes on moderate loading (75% of max. heart rate), 5 minutes cool down. Strengthening Exercises Conventional Exercise Program: 2 times per week for 4 weeks Heat Therapy Ultrasound Therapy
  * Static Quadriceps activation 10*2 RM
  * SLR 10*2 RM
  * VMO activation 10*2 RM
  * Knee to Chest 5*2 RM
  * Quads, Hams & Calf stretches
  Interventions: Other: Group B will receive aerobic and strength training and conventional physiotherapy protocol for knee OA only.

INTERVENTIONS:
Other: Group A will receive Voodoo Flossing Technique along with aerobic and strengthening exercises & conventional physiotherapy protocol for Knee OA. — Patient will sit or lie down comfortably with affected knee exposed and in extension. Start by wrapping voodoo floss band at the shin bone just below the knee joint with 50% tension in the band and 50% overlapping on each wrap by working your way up towards the thigh. Keep the flossing band on for at least 1-2 minutes and perform gentle knee movements to promote mobility.
  * Knee flexion and extension in full range of motion in standing position 20-30 sec.
  * Knee squats with/without support 20-30 sec.
  * Abduction and Adduction 20-30 sec. Perform each exercise with 10-15 seconds of rest between each set. After completing ROM exercises, allow the knee to rest in comfortable position and then carefully unwrap the voodoo band from the knee joint. Also monitor the knee for any changes.
  Arms: Voodoo Flossing technique along with aerobic & strengthening exercises and conventional protocol.
Other: Group B will receive aerobic and strength training and conventional physiotherapy protocol for knee OA only. — Aerobic Exercises: Walking or Stationary Cycling 2 times a week for 4 weeks Walking: On flat surface/Treadmill
  * 10 minutes warm-up, 30 minutes brisk walking, 5 minutes cool down. Cycling: Ergometer cycling
  * 10 minutes warm-up, 30 minutes on moderate loading (75% of max. heart rate), 5 minutes cool down. Strengthening Exercises: Quadriceps, Hamstrings, Hip Abductors, Adductors and Calf Muscles Strengthening and Balance Training 2 times a week for 4 weeks.
  * Hip Abduction in standing 8-10*2 RM
  * Hip Adduction in standing 8-10*2 RM
  * Knee Flexion and Extension in standing 10*2 RM
  * Knee Squats 8-10*2 RM
  * Sit/stand from chair 10*2 RM
  * Step up and down 10*2 RM
  * Heel raises 10*2 RM
  * Hip Bridges 10*2 RM Conventional Exercise Program: 2 times per week for 4 weeks Heat Therapy Ultrasound Therapy
  * Static Quads activation 10*2 RM
  * SLR 10*2 RM
  * VMO activation 10*2 RM
  * Knee to Chest 5*2 RM
  * Quadriceps, Hamstrings and Calf stretches 5*2 RM
  Arms: Aerobic and strength training and conventional physiotherapy protocol for knee OA.

SUMMARY:
Knee osteoarthritis (KOA) is a prevalent degenerative joint disease characterized by pain, stiffness, and reduced physical function, significantly impacting quality of life especially in elderly population. This study aims to evaluating the effectiveness of an emerging technique, known as 'Voodoo Flossing' on pain, range of motion and physical function in KOA to provide evidence-based insight of voodoo flossing as a potential therapeutic adjunct in KOA management.

This randomized controlled trial will be conducted at Riphah Rehabilitation Clinic, Lahore and Horizon Hospital Lahore in a time span of 8 months. A sample size of 42 subjects selected through non-probability convenient sampling with age group between 45 to 65 having present complain confirmed through Kellgren-Lawrence (KL) scale of grade-II will be divided into two groups, will undergo aerobic exercises, strengthening exercises and conventional physiotherapy protocol either with or without Voodoo Flossing technique.

DETAILED DESCRIPTION:
A double blinded randomized controlled trial has been conducted to investigate the effectiveness of integrating flossing band therapy with conventional physiotherapy, anticipating outcomes of pain reduction, functional ability, and patient satisfaction. Outcomes were measured for pain (VAS), strength (Dynamometry), lower limb function (LEFS) and PFPS function (AKPS) before and after intervention stating flossing band integrated with physiotherapy as more effective treatment modality for PFPS.

A study has been conducted to check the effectiveness of voodoo flossing on pain and functional recovery in shin splint on amateur runners. Pre and post-test measurements were taken showing voodoo flossing as an effective technique for reducing pain and improving pain free activities in management of Shin Splint Syndrome in amateur runners.

A randomized control trial aimed to compare the lasting effects of the flossing band (FB) technique, dynamic stretching (DS) and static stretching (SS) on hamstring, on knee ROM, muscle activity, and proprioception to identify the most effective pre-exercise method for preventing injuries. FB group shows improvements in joint ROM and muscle activity as compared to DS and SS groups and exhibited lasting effects. Also, the proprioception observed at 30°, 60°, and 90° knee flexion had the smallest repositioning error in the FB group. Previous researches have shown positive aspects of voodoo flossing combined with physiotherapy on ankle joint, shoulder joint, shin splints, PFPS, knee ROM, proprioception, muscle functionality but evidence of its application in knee OA patients is scarce. By systematically addressing these gaps through well designed RCTs and comprehensive outcome assessments, future research can provide evidence-based insight of voodoo flossing as a potential therapeutic adjunct in KOA management. This study aims to address this existing literature gap by elucidating its potential effects on knee pain, ROM and physical function in KOA patients and making future recommendations for further study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 45 and ≤ 65
* Both Male and Female
* Knee Pain persisting for at-least 3 months
* Pain severity during walking ≥ 2/10 on a Numeric Pain Rating Scale
* Walking and Balance (Mobility) problems according to Time Up & Go (TUG) test
* Poor scoring on WOMAC scale for pain, stiffness and physical activities
* Knee OA Grade II (according to Kellgren-Lawrence method)
* Participants must provide informed consent for participation in RCT

Exclusion Criteria:

* Age < 45 and > 65
* Severe Knee pain during Walking ≥ 9/10 on a Numeric Pain Rating Scale
* Knee OA Grade I, III & IV (according to Kellgren-Lawrence method)
* Physical or Mental co-morbidity severely affecting daily life of patient
* Any Contraindication to provide Exercise Therapy
* Suspicion of chronic widespread pain (i.e., pain present for at least 3 months in at least three joints including left and right side of the body, above and below the waist, and the axial skeleton)
* Participant undergone total knee arthroplasty or on waiting list for total knee arthroplasty in any knee
* Any other reasons for knee pain than knee OA (e.g., rheumatoid arthritis and gout)
* Received intraarticular injections in past 6 months because of knee pain (Hyaluronic Gel or steroid)

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 4th week
  Patient level of pain will be assessed using this scale. This scale ranges from 0 to 10. 0 indicates "no pain" and 10 indicates "worst pain". In this study, participants rating ≥2 and ≤9 on NPRS will be taken.
The Western Ontario and McMaster Universities Osteoarthritis Index | 4th week
  WOMAC index is a widely used questionnaire designed to assess the three dimensions of pain, stiffness, and physical function in individuals with OA of the hip or knee. It is a 24-item questionnaire divided into three sub-categories: Pain (5 items), Stiffness (2 items), Physical Function (17 items). Participants having poor scoring on WOMAC scale for pain, stiffness and physical activities will be considered for this study.

SECONDARY OUTCOMES:
Time Up & Go Test | 4th week
  Time Up and Go (TUG) test is a simple, quick, and reliable clinical tool used to assess functional mobility, balance, and gait speed by measuring the time it takes for an individual to rise from a chair (or seated position), walk a short distance (typically 3 meters or 10 feet), turn around, walk back to the chair, and sit down again. A score of ≤ 14 seconds has been shown to indicate high risk of falls.
Universal Goniometer | 4th week
  The range of motion will be measured by using Universal Goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Hira Shaukat, TDPT, Principal Investigator — Riphah International University
Locations (1):
- Horizon Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Acar S, Aljumaa H, Sevik K, Karatosun V, Unver B. The Intrarater and Interrater Reliability and Validity of Universal Goniometer, Digital Inclinometer, and Smartphone Application Measuring Range of Motion in Patients with Total Knee Arthroplasty. Indian J Orthop. 2024 Apr 19;58(6):732-739. doi: 10.1007/s43465-024-01129-z. eCollection 2024 Jun. PMID 38812867
- [Background] Oiestad BE, Aroen A, Rotterud JH, Osteras N, Jarstad E, Grotle M, Risberg MA. The efficacy of strength or aerobic exercise on quality of life and knee function in patients with knee osteoarthritis. A multi-arm randomized controlled trial with 1-year follow-up. BMC Musculoskelet Disord. 2023 Sep 8;24(1):714. doi: 10.1186/s12891-023-06831-x. PMID 37684597
- [Background] Kelly CF, Oliveri Z, Saladino J, Senatore J, Kamat A, Zarour J, Douris PC. The Acute Effect of Tissue Flossing on Pain, Function, and Perception of Movement: A Pilot Study. Int J Exerc Sci. 2023 Jul 1;16(3):855-865. doi: 10.70252/OKAO5505. eCollection 2023. PMID 37637031
- [Background] Tore NG, Oskay D, Haznedaroglu S. The quality of physiotherapy and rehabilitation program and the effect of telerehabilitation on patients with knee osteoarthritis. Clin Rheumatol. 2023 Mar;42(3):903-915. doi: 10.1007/s10067-022-06417-3. Epub 2022 Oct 24. PMID 36279075
- [Background] Geng R, Li J, Yu C, Zhang C, Chen F, Chen J, Ni H, Wang J, Kang K, Wei Z, Xu Y, Jin T. Knee osteoarthritis: Current status and research progress in treatment (Review). Exp Ther Med. 2023 Aug 25;26(4):481. doi: 10.3892/etm.2023.12180. eCollection 2023 Oct. PMID 37745043